CLINICAL TRIAL: NCT03973411
Title: Ondansetron in the Prevention of Hypotension in Patients Undergoing Spinal Anesthesia: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Ondansetron in the Prevention of Hypotension in Patients Undergoing Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Preceptor of medical residency in anesthesiology, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ondansetron for spinal
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Hypotension
Keywords: Ondansetron; Hypotension; Spinal anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, duble-blind and placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron group (Active Comparator): Patients will receive intravenous ondansetron before spinal anesthesia
  Interventions: Drug: Prophylactic ondansetron
- Control group (Placebo Comparator): Patients will receive intravenous saline before spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prophylactic ondansetron — Pacients will receibe prophylactic ondansetron plus standard spinal anesthesia
  Arms: Ondansetron group
Drug: Placebo — Pacients will receibe standard spinal anesthesia
  Arms: Control group

SUMMARY:
Ondansetron, a potent 5-HT 3 receptor antagonist commonly used as an antiemetic. The main objective of the present study is to verify the hypothesis that blocking type 3 serotonin receptors with intravenous ondansetron reduces the incidence of spinal anesthesia-induced hypotension

DETAILED DESCRIPTION:
Spinal anesthesia is usually the first choice for many surgical procedures of lower limbs, perineum, and lower abdomen. It is a simple and safe procedure, however it can present complications such as hypotension and bradycardia.

Hypotension results mainly from a decrease in systemic vascular resistance secondary to a blockage of sympathetic fibers. The Bezold-Jarisch reflex, proposed as a mechanism for bradycardia is mediated by serotonin receptors (subtype 5-HT3) located in the vagus nerve and within the walls of the cardiac ventricles. 5-HT3 receptors are activated in response to systemic hypotension, causing increased vagal efferent signaling, bradycardia, reduced cardiac output and increased exacerbation of hypotension.

Therefore, ondansetron, a potent 5-HT 3 receptor antagonist commonly used as an antiemetic, is potentially useful in attenuating this response. To assess this response, the main goal of the present study is to verify the hypothesis that blocking type 3 serotonin receptors with intravenous ondansetron reduces the incidence of spinal anesthesia-induced hypotension.

This prospective, randomized, double-blind, placebo-controlled study aims to verify the hypothesis that blocking serotonin type 3 receptors with intravenous ondansetron prior to subarachnoid block reduces hypotension induced by spinal anesthesia in surgical procedures at Base Hospital of the Federal District. The examiners responsible for patient assessment will not have access to the agents used.

Patients will be randomized through a randomly generated list. The examiner responsible for opening the envelope will make the draw, will include the patient in one of the groups, write down their data in the random list, prepare the syringe with the medication, and deliver it to the operating room so that the next examiners will not be aware of the administered drug.

Patients will receive standard monitoring, venoclysis, intravenous midazolam as pre-anesthetic medication. The study drug (ondansetron 0.15 mg / kg or placebo) will then be administered. All patients received spinal anesthesia with hyperbaric bupivacaine and opioid adjuvants at the discretion of the anesthesiologist.

The evolution of vital signs such as systolic blood pressure, mean heart rate, height of the sensitive block, incidence of adverse events such as bradycardia, tachycardia, hypertension or hypotension, nausea, vomiting, vasopressor and antiemetic consumption will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years, electively scaled for surgery requiring neuraxial block, with programming of spinal anesthesia.
* Physical State 1, 2 or 3 of the American Society of Anesthesiology (ASA)

Exclusion Criteria:

* Patients taking prophylactic or therapeutic anticoagulation, except respecting the allowed range;
* Patients with atrioventricular block
* Patients with cardiac arrhythmias
* Patients with heart failure;
* Patients with renal disease
* Patients with liver disease
* Patient carrying or suspecting any type of systemic infection or located in a puncture site;
* Patients who refuse to participate in the study after presenting the free and informed consent form;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as hypotension | During surgery
  Intraoperative hemodynamic stability analysis through the incidence bradycardia, hypotension and consumed vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonça, MD, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil